CLINICAL TRIAL: NCT01277510
Title: A Randomized, Double-blind, Placebo Controlled Study to Assess the Efficacy and Safety of Cinacalcet HCl in Pediatric Subjects With Chronic Kidney Disease and Secondary Hyperparathyroidism Receiving Dialysis
Brief Title: Pediatric Chronic Kidney Disease Safety and Efficacy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was put on clinical hold on 30 Jan 2013 following a subject fatality. Study was never restarted and was closed.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20070208
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Chronic Kidney Disease; Hyperparathyroidism; Hyperparathyroidism, Secondary; Kidney Disease; Secondary Hyperparathyroidism
Keywords: dialysis; sensipar; mimpara; hemodialysis; peritoneal dialysis; renal; parathyroid hormone; pediatric
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism; Hyperparathyroidism, Secondary; Kidney Diseases | interventions — Cinacalcet; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received standard of care and placebo once daily for 30 weeks during the double-blind phase. During the open-label phase, participants received cinacalcet with standard of care for an additional 30 weeks. The starting dose of cinacalcet was ≤ 0.20 mg/kg based on dry weight, and could be titrated up according to plasma iPTH and serum calcium levels every 4 weeks up to Week 54 to a maximum dose of 4.2 mg/kg.
  Interventions: Drug: placebo; Drug: Standard of Care
- Cinacalcet (Experimental): Participants received standard of care and cinacalcet once daily for 30 weeks during the double-blind phase. The starting dose of cinacalcet was ≤ 0.20 mg/kg based on dry weight, and could be titrated up according to plasma iPTH and serum calcium levels every 4 weeks until Week 24 to a maximum dose of 4.2 mg/kg. During the open-label phase participants continued to receive cinacalcet with standard of care for an additional 30 weeks.
  Interventions: Drug: cinacalcet capsule; Drug: Standard of Care

INTERVENTIONS:
Drug: cinacalcet capsule — Cinacalcet was prepared for oral administration as both capsules for sprinkling and film coated tablets for swallowing.
  Other Names: Sensipar, Mimpara
  Arms: Cinacalcet
Drug: placebo — Placebo tablets and capsules for sprinkling identical to active treatment.
  Arms: Placebo
Drug: Standard of Care — All participants, regardless of treatment assignment, will receive standard of care with vitamin D sterols (calcitriol and its analogs), as prescribed by the treating physician.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of adding cinacalcet to the current treatment of secondary hyperparathyroidism in children currently receiving dialysis compared to a treatment regimen that does not include cinacalcet.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism (SHPT) is a condition that can develop early in patients with chronic kidney disease (CKD), usually gets worse over time, and is known to cause problems for patients on dialysis. Children on dialysis can have a wide range of bone and growth issues, and common treatments have a chance of making these things worse by increasing serum calcium and serum phosphorus. Cinacalcet has been shown to be effective in controlling parathyroid hormone (PTH), calcium and phosphorus in adults. The purpose of this study is to show that including cinacalcet in the treatment of SHPT will lower the levels of intact parathyroid hormone (iPTH) in a larger number of pediatric patients with CKD who are receiving dialysis, compared to a treatment regimen that does not include cinacalcet.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to less than 18 years at screening
* Diagnosed with CKD and SHPT receiving hemodialysis or peritoneal dialysis for ≥ 2 months before randomization
* Dry weight ≥ 12.5 kg at screening
* iPTH obtained from the central laboratory must be > 300 pg/mL (31.8 pmol/L)
* Serum calcium (corrected) obtained from the central laboratory must be ≥ 8.8 mg/dL (2.2 mmol/L)
* Serum phosphorus obtained from the central laboratory ≥ 4.0 mg/dL (1.3 mmol/L) for children 6 to less than 12 years old, or ≥ 3.5 mg/dL (1.1 mmol/L) for children 12 to less than 18 years old
* Subjects already receiving vitamin D sterols (either calcitriol or a synthetic analog), a stable dose within the last 2 months prior to randomization
* Subjects taking growth hormone, a stable dose defined as no change > than 20% in the last 2 months prior to randomization
* Subjects on anti-convulsant medication must be on a stable dose for 3 months, and have a therapeutic blood level of the anti-convulsant at the time of randomization
* Subjects must be on a dialysate calcium concentration of ≥ 2.5 mEq/L (1.25 mmol/L) for at least 2 months prior to randomization

Exclusion Criteria:

* Underwent parathyroidectomy in the last 6 months
* Anticipated parathyroidectomy within 6 months after randomization
* Received therapy with cinacalcet (sensipar/mimpara) within the last month
* A new onset of seizure or worsening of a pre-existing seizure disorder within the last 3 months
* Scheduled date for kidney transplant from a known living donor that makes completion of the study unlikely

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2014-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (49):
- United States (17):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Gainesville, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Livingston, New Jersey
  - Research Site, The Bronx, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
- Australia (4):
  - Research Site, Randwick, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Parkville, Victoria
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
- Germany (2):
  - Research Site, Heidelberg
  - Research Site, Marburg
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
  - Research Site, Szeged
- Mexico (2):
  - Research Site, Mexico City, Mexico City
  - Research Site, Aguascalientes
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Gorzów Wielkopolski
  - Research Site, Lodz
  - Research Site, Warsaw
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Samara
- Slovakia (3):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
- Spain (6):
  - Research Site, Barakaldo, Basque Country
  - Research Site, Barcelona, Catalonia
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, Barakaldo, PaÃ-s Vasco
  - Research Site, Valencia, Valencia
  - Research Site, Madrid

REFERENCES:
- [Background] Warady BA, Iles JN, Ariceta G, Dehmel B, Hidalgo G, Jiang X, Laskin B, Shahinfar S, Vande Walle J, Schaefer F. A randomized, double-blind, placebo-controlled study to assess the efficacy and safety of cinacalcet in pediatric patients with chronic kidney disease and secondary hyperparathyroidism receiving dialysis. Pediatr Nephrol. 2019 Mar;34(3):475-486. doi: 10.1007/s00467-018-4116-y. Epub 2018 Nov 30. PMID 30506144
- [Background] Warady BA, Ng E, Bloss L, Mo M, Schaefer F, Bacchetta J. Cinacalcet studies in pediatric subjects with secondary hyperparathyroidism receiving dialysis. Pediatr Nephrol. 2020 Sep;35(9):1679-1697. doi: 10.1007/s00467-020-04516-4. Epub 2020 May 4. PMID 32367309
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 28 June 2011 and the last patient enrolled was on 15 January 2013.
  Eligible participants were between the ages of 6 to less than 18 years old who had chronic kidney (CKD) and secondary hyperparathyroidism treated with either hemodialysis or peritoneal dialysis for ≥ 2 months.
Pre-assignment Details: This study consisted of a 30-week randomized, double-blind phase followed by a 30-week open-label phase. Participants were randomized 1:1 to receive either cinacalcet or placebo in the double-blind phase. All participants received cinacalcet in the open-label phase.
Groups:
- Cinacalcet: Participants received standard of care and cinacalcet once daily for 30 weeks during the double-blind phase. The starting dose of cinacalcet was ≤ 0.20 mg/kg based on dry weight, and could be titrated up according to plasma iPTH and serum calcium levels every 4 weeks until Week 24 to a maximum dose of 4.2 mg/kg. During the open-label phase participants continued to receive cinacalcet with standard of care for an additional 30 weeks. Regardless of the titration level reached at the last dose of IP in the double-blind phase, all participants started titration at ≤ 0.20 mg/kg based on dry weight.
Period: Double-blind Phase
Arm/Group | Placebo | Cinacalcet
Started | 21 | 22
Received Investigational Product | 21 | 22
Completed | 8 (Completed investigational product) | 4 (Completed investigational product)
Not Completed | 13 | 18
Not completed — Non-compliance | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Administrative decision | 7 | 9
Not completed — Death | 0 | 1
Not completed — Protocol-specified criteria | 2 | 6
Not completed — Other | 1 | 1
Period: Open-label Phase
Arm/Group | Placebo | Cinacalcet
Started | 8 | 4
Received Investigational Product | 6 | 4
Completed | 1 (Completed investigational product) | 1 (Completed investigational product)
Not Completed | 7 | 3
Not completed — Administrative decision | 4 | 3
Not completed — Protocol-specified criteria | 1 | 0
Not completed — Never received investigational product | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cinacalcet | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (2.9) | 13.3 (3.6) | 13.2 (3.3)
Age, Customized [Number; unit: participants]
  6 to < 12 years | 5 | 6 | 11
  12 to < 18 years | 16 | 16 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Number; unit: participants]
  White | 15 | 16 | 31
  Black or African American | 6 | 5 | 11
  Other | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 16 | 19 | 35
Intact Parathyroid Hormone (iPTH) [Mean (Standard Deviation); unit: pg/mL] | 795.8 (537.9) | 757.1 (440.1) | 776.0 (484.8)
Corrected Total Serum Calcium [Mean (Standard Deviation); unit: mg/dL] — Serum calcium was reported as a corrected value by the central laboratory based on calcium and albumin concentrations:
  Corrected total calcium (mg/dL) = measured total serum calcium (mg/dL) + 0.8 (4.0 - Serum albumin (g/dL)).
  mg/dL | 9.88 (0.62) | 9.91 (0.54) | 9.90 (0.58)
Serum Phosphorous [Mean (Standard Deviation); unit: mg/dL] | 6.37 (1.48) | 6.68 (1.78) | 6.53 (1.63)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ≥ 30% Reduction in Mean iPTH From Baseline to the Efficacy Assessment Phase
Description: The efficacy assessment value is based on the scheduled assessment(s) taken during the efficacy assessment phase (EAP; Weeks 25 - 30). When multiple assessments were available, the average of those was used. If an efficacy measurement during the EAP was missing, the mean of the last 2 available post-baseline values in the dose-titration phase was used. If only one post-baseline value was available, this single value was used.
Time Frame: From Baseline to the Efficacy Assessment Phase, Weeks 25-30
Population: Full analysis set, which includes all randomized participants with at least 1 post-baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 21 | 22
percentage of participants | 19.0 | 54.5
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; A hierarchical testing procedure was used to test the primary and biochemical secondary endpoints (Outcome Measures 1-5). The primary endpoint was tested at a significance level of 0.05. The four biochemical secondary endpoints were to be tested using Holm's method at 0.05 should the primary endpoint achieve a significant result; Test type: Superiority or Other; p = 0.017, Cochran-Mantel-Haenszel; Cochran- Mantel-Haenszel (CMH) test stratified by baseline age group (6 -<12 years old or 12 - <18 years old); Difference (Cinacalcet - Placebo) = 35.50, 95% CI 2-sided [8.76 to 62.24]

2. Secondary Outcome: Percentage of Participants Achieving Mean iPTH ≤ 300 pg/mL (31.8 Pmol/L) During the Efficacy Assessment Phase
Description: The efficacy assessment value is based on the scheduled assessment(s) taken during the efficacy assessment phase. When multiple assessments were available, the average of those was used. If an efficacy measurement during the EAP was missing, the mean of the last 2 available postbaseline values in the dose-titration phase was used. If only one post-baseline value was available, this single value was used.
Time Frame: From Baseline to the Efficacy Assessment Phase (EAP), Weeks 25-30
Population: Full analysis set
Measure: Number; unit: pecentage of participants
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 21 | 22
pecentage of participants | 23.8 | 27.3
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; The secondary endpoint with the smallest p-value was first compared at a significance level of 0.0125. If the p-value was > 0.0125, all 4 secondary endpoints were non-significant; if ≤ 0.0125, the null hypothesis for that endpoint was rejected. Next, the 2nd smallest p-value was compared at a level of 0.0167; if > 0.0167, the remaining 3 endpoints were not significant, or, the null hypothesis of that endpoint was rejected. The other 2 endpoints were analyzed similarly, at 0.025 and 0.05; Test type: Superiority or Other; p = 0.826, Cochran-Mantel-Haenszel; Cochran- Mantel-Haenszel (CMH) test stratified by baseline age group (6 -<12 years old or 12 - <18 years old); Difference (Cinacalcet - Placebo) = 3.46, 95% CI 2-sided [-22.58 to 29.51]

3. Secondary Outcome: Percent Change From Baseline in Mean Corrected Total Serum Calcium During the Efficacy Assessment Period
Description: Serum calcium was reported as a corrected value by the central laboratory based on calcium and albumin concentrations: Corrected total calcium (mg/dL) = measured total serum calcium (mg/dL) + 0.8 (4.0 - Serum albumin (g/dL)). The efficacy assessment value is based on the scheduled assessment(s) taken during the efficacy assessment phase. When multiple assessments were available, the average of those was used. If an efficacy measurement during the EAP was missing, the mean of the last 2 available postbaseline values in the dose-titration phase was used. If only one post-baseline value was available, this single value was used."
Time Frame: From Baseline to the Efficacy Assessment Phase, Weeks 25-30.
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 21 | 22
percent change | -1.0 (1.91) [-4.9 to 2.9] | -4.6 (1.84) [-8.4 to -0.9]
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.147, ANCOVA; Baseline age group was used as covariate; LS Mean Difference = -3.7, 95% CI 2-sided [-8.6 to 1.3] — Cinacalcet-Placebo

4. Secondary Outcome: Percent Change From Baseline in Mean Serum Phosphorus During the Efficacy Assessment Phase
Description: as for outcome 2
Time Frame: From Baseline to the Efficacy Assessment Phase, Weeks 25-30.
Population: Full analysis set; data for one participant in the Placebo group were not available.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 20 | 22
percent change | 10.2 [-0.8 to 21.2] | 4.9 [-5.5 to 15.3]
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.454, ANCOVA; Baseline age group was used as covariate; LS Mean Difference = -5.3, 95% CI 2-sided [-19.4 to 8.9] — Cinacalcet-Placebo

5. Secondary Outcome: Percent Change From Baseline in Mean Phosphorous Product (Ca x P) During the Efficacy Assessment Phase
Description: as for outcome 2
Time Frame: From Baseline to end of Efficacy Assessment Period, assessed up to 30 weeks
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 21 | 22
percent change | 8.0 [-1.8 to 17.7] | -2.0 [-11.4 to 7.4]
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.117, ANCOVA; Baseline age group was used as covariate; LS Mean Difference = -10.0, 95% CI 2-sided [-22.5 to 2.6] — Cinacalcet-Placebo

6. Secondary Outcome: Growth Velocity From Baseline to End of Double-blind Phase
Description: Linear growth velocity (cm/year) = 52 x change in height (cm) / number of weeks between the two assessments. End of double-blind phase visit was at Week 30 by design but the last assessment in the double-blind phase was used due to the early termination of the study.
Time Frame: From Baseline to end of Efficacy Assessment at Week 30
Population: Full analysis set; the last assessment in the double-blind phase was used due to the early termination of the study. Only participants with available data are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/year
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 19 | 17
cm/year | 3.1 [0.7 to 5.6] | 3.3 [0.8 to 5.8]
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p = 0.896, ANCOVA — No adjustments for multiplicity were made; Baseline age group was used as covariate; LS Mean Difference = 0.2, 95% CI 2-sided [-3.1 to 3.6] — Cinacalcet-Placebo

7. Secondary Outcome: Growth Velocity From End of Double-blind Phase to End of Open-label Phase
Description: Linear growth velocity (cm/year) = 52 x change in height (cm) / number of weeks between the two assessments. End of open-label phase visit was at Week 60 by design but the last assessment in the open-label phase was used due to the early termination of the study.
Time Frame: End of double-blind phase (Week 30) until end of the open-label phase (Week 60)
Population: Full analysis set. Only participants with available data were included in the anaysis.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 7 | 3
cm/year | 2.75 (3.23) | 1.21 (1.31)

8. Secondary Outcome: Percent Change From Baseline in Mean Ionized Calcium During the Efficacy Assessment Phase
Description: as for outcome 2
Time Frame: From Baseline to the Efficacy Assessment Phase, Weeks 25-30.
Population: Full analysis set; only participants with available data were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 12 | 18
percent change | -1.5 [-8.6 to 5.6] | -2.3 [-8.2 to 3.5]
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p = 0.854, ANCOVA; Baseline age group was used as covariate; LS Mean Difference = -0.8, 95% CI 2-sided [-9.4 to 7.9] — Cinacalcet-Placebo

ADVERSE EVENTS:
Time Frame: 60 Weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Cinacalcet | Open-label Phase: Previous Placebo | Open-label Phase: Previous Cinacalcet
Serious Adverse Events (participants affected / at risk) | 9/21 | 9/22 | 3/6 | 1/4
Other Adverse Events (participants affected / at risk) | 17/21 | 16/22 | 6/6 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: Placebo (N=21) | Double-blind Phase: Cinacalcet (N=22) | Open-label Phase: Previous Placebo (N=6) | Open-label Phase: Previous Cinacalcet (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Papilloedema (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Medical device complication (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0
Thrombosis in device (General disorders) | 0 | 1 | 0 | 0
Rubber sensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Transplant rejection (Immune system disorders) | 1 | 0 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Measles (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: Placebo (N=21) | Double-blind Phase: Cinacalcet (N=22) | Open-label Phase: Previous Placebo (N=6) | Open-label Phase: Previous Cinacalcet (N=4)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 7 | 1 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0
Catheter site pruritus (General disorders) | 0 | 1 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 2 | 1 | 1 | 0
Device breakage (General disorders) | 1 | 0 | 0 | 0
Device leakage (General disorders) | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 0 | 0
Local swelling (General disorders) | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 2 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dialysis related complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood calcium abnormal (Investigations) | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 5 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 3 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0
Daydreaming (Psychiatric disorders) | 0 | 1 | 0 | 0
Staring (Psychiatric disorders) | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early with a smaller sample size. However, the study was still sufficiently powered for the double-blind phase. The data collected in the open-label phase is very sparse.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.